CLINICAL TRIAL: NCT02427347
Title: A Randomized Controlled Clinical Trial of Acupuncture on Regulating Dai Meridian for Visceral Fat Metabolism in Abdominal Obesity.
Brief Title: Acupuncture in the Regulation of Dai Meridian for the Metabolism of Visceral Adipose Tissue in Abdominal Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dongfang Hospital Beijing University of Chinese Medicine (Other)
Collaborators: Beijing Municipal Science & Technology Commission (Other); Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Hui Hu, Principal Investigator, Dongfang Hospital Beijing University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Z141107002514079
Record Dates: First submitted 2015-04-13; First posted 2015-04-28 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Abdominal Obesity; Metabolic Syndrome
MeSH Terms: conditions — Obesity, Abdominal; Metabolic Syndrome | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Intervention including acupuncture treatment and healthy education.
  Interventions: Other: Acupuncture; Other: Healthy education
- Control group (Other): Healthy education is given as a baseline treatment.
  Interventions: Other: Healthy education

INTERVENTIONS:
Other: Acupuncture — Acupuncture needles of 0.3mm in diameter and 100mm in length are inserted into gallbladder-meridian(GB)26 about 25-65mm deep by an angle of 15°, following the path of Dai Meridian (towards medial and downside) . The other acupoints are inserted with needles of 0.25-0.3mm in diameter and 25-40mm in length approximately 10-30mm deep, with an angle of 90°. Electro-acupuncture is applied to both sides of GB26 and stomach-meridian(ST)25: cathode is connected to GB26; anode to ST25. Dense-disperse wave pattern and a wave frequency of 2/100 Hertz is chosen. The intensity of the electro-acupuncture is adjusted on average 4-8 milliampere. The needles are subsequently retained for 20min. The results of the study are based on 8 weeks, each week consisting of 3 sessions.
  Arms: Intervention group
Other: Healthy education — Healthy knowledge lectures and issuing brochures are given. Education of patients for conditioning and changing bad habits, diet, quit smoking, limit alcohol consumption, salt restriction, appropriate increase in physical activity.

SUMMARY:
To evaluate the effectiveness of acupuncture therapy combined with healthy education for patients with abdominal obesity.

DETAILED DESCRIPTION:
This subject is a prospective, single-blind, parallel-group, randomized controlled clinical trial.120 patients with abdominal obesity are allocated into two groups with a ratio of 2:1.Randomized series was generated by computer. The allocation was concealed. Patients in the intervention group are received acupuncture therapy and healthy education. Patients in the control group are only given healthy education. The treatment in both intervention group and control group lasts for 8 weeks. Comparison of two groups of patients with abdominal fat thickness, fasting serum visfatin concentration, simple anthropometric parameters (including body weight, body mass index, waist circumference, hip circumference, waist-to-hip radio, waist-to-height radio, the percentage of body fat), fasting blood glucose, fasting insulin, glycosylated hemoglobin, fasting blood lipid (total cholesterol, triglyceride, high density lipoprotein, low density lipoprotein), uric acid, blood pressure, insulin resistance level, and obesity related lifestyle survey.

ELIGIBILITY:
Inclusion Criteria:

* Met the diagnostic criteria of abdominal obesity (waist circumference of male ≥ 90cm, waist circumference of female ≥ 80cm);
* Ultrasound viscerofatty index ≥ 3;
* Age between 18-70 years old;
* Signed informed consent voluntarily.

Exclusion Criteria:

* Secondary obesity caused by endocrine, hereditary, nervous system,or drugs;
* Within 3 months adjusted drug therapy for diabetes or hypertension or hyperlipidemia;
* undergoing other therapies for reducing body mass and waist circumference, such as surgery, medication, etc;
* participating or have participated in other studies;
* pregnant or breast-feeding women;
* critically ill, having hepatic-renal dysfunction or mental illness;
* severe impairment in sight and hearing.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline in abdominal subcutaneous fat thickness at 8 weeks | baseline and 8 weeks
  Including subcutaneous fat thickness 1 and 2
Changes from Baseline in abdominal visceral fat thickness at 8 weeks | baseline and 8 weeks
  Including visceral fat thickness 1 and 2
Change from Baseline in antero-hepatic fat thickness at 8 weeks | baseline and 8 weeks
  Antero-hepatic fat thickness (AHF) was determined by the distance of peritoneum to the hepatic cortex at the subcostal level.
Change from Baseline in perirenal fat thickness at 8 weeks | baseline and 8 weeks
  Perirenal fat thickness (PRF) was determined by the thickest one of the perirenal fat capsule of the right kidney short axis, when the right renal short axis and the maximum width of the renal sinus were clearly displayed.
Change from Baseline in ultrasound viscerofatty index at 8 weeks | baseline and 8 weeks
  ultrasound viscerofatty index (UVI) = (visceral fat thickness 1 + visceral fat thickness2)/(subcutaneous fat thickness 1 + subcutaneous fat thickness 2)
Change from Baseline in fasting serum visfatin at 8 weeks | baseline and 8 weeks
  5ml venous blood was told after an 8 hours fast. Visfatin was measured by enzyme-linkedimmuno sorbent assay (ELISA).

SECONDARY OUTCOMES:
Change from Baseline in body weight | baseline, 4 weeks and 8 weeks
  It's made at the situation of fasting, after emptying bowels, with minimal clothing, without headdress and footwear, at the end of expiration.
Change from Baseline in body mass index | baseline, 4 weeks and 8 weeks
  Body mass index (BMI) = body weight(kg)/height(m)/height(m)
Change from Baseline in waist circumference | baseline, 4 weeks and 8 weeks
  WC was measured at the level between the inferior portion of 12th rib and iliac crest.
Change from Baseline in hip circumference | baseline, 4 weeks and 8 weeks
  HC was measured at the level of the most prominent point of the pelvis.
Change from Baseline in waist-to-hip radio | baseline, 4 weeks and 8 weeks
  waist-to-hip radio (WHR) = waist circumference(cm)/hip circumference(cm)
Change from Baseline in waist-to-height radio | baseline, 4 weeks and 8 weeks
  waist-to-height radio (WHtR) = waist circumference(cm)/height(cm)
Change from Baseline in the percentage of body fat | baseline, 4 weeks and 8 weeks
  the percentage of body fat = 1.2×BMI+0.23×age-5.4-10.8×gender（M=1，F=0）
Change from Baseline in fasting blood glucose at 8 weeks | baseline and 8 weeks
  5ml venous blood was collected after an 8 hours fast. It was tested by our hospital's laboratory.
Change from Baseline in fasting insulin at 8 weeks | baseline and 8 weeks
  5ml venous blood was collected after an 8 hours fast. It was tested by our hospital's laboratory.
Change from Baseline in glycosylated hemoglobin at 8 weeks | baseline and 8 weeks
  5ml venous blood was collected after an 8 hours fast. It was tested by our hospital's laboratory.
Change from Baseline in fasting total cholesterol at 8 weeks | baseline and 8 weeks
  5ml venous blood was collected after an 8 hours fast. It was tested by our hospital's laboratory.
Change from Baseline in fasting triglyceride at 8 weeks | baseline and 8 weeks
  5ml venous blood was collected after an 8 hours fast. It was tested by our hospital's laboratory.
Change from Baseline in fasting high density lipoprotein cholesterol at 8 weeks | baseline and 8 weeks
  5ml venous blood was collected after an 8 hours fast. It was tested by our hospital's laboratory.
Change from Baseline in fasting low density lipoprotein cholesterol at 8 weeks | baseline and 8 weeks
  5ml venous blood was collected after an 8 hours fast. It was tested by our hospital's laboratory.
Change from Baseline in fasting uric acid at 8 weeks | baseline and 8 weeks
  5ml venous blood was collected after an 8 hours fast. It was tested by our hospital's laboratory.
Change from Baseline in blood pressure at 8 weeks | baseline and 8 weeks
Change from Baseline in insulin resistance level at 8 weeks | baseline and 8 weeks
Change from Baseline in obesity related lifestyle survey at 8 weeks | baseline and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hui Hu, doctor, Study Chair — Department of Acupuncture and Moxibustion, Dongfang Hospital, Beijing University of Chinese Medicine
Locations (1):
- Department of Acupuncture and Moxibustion, Dongfang Hospital, Beijing University of Chinese Medicine, Beijing, Beijing Municipality, China